CLINICAL TRIAL: NCT05685043
Title: Clinical Outcome and Cost Following a CT-perfusion Imaging Decision for Mechanical Thrombectomy in Acute Ischaemic Stroke Within the Time Window of 6 Hours: a Randomised, Controlled, Partially Blinded Multicenter Non-inferiority Study
Brief Title: BELgian CT-perFUSion Study to Select Acute Stroke Patients for Thrombectomy
Acronym: BELFUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding available.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-11282
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic
Keywords: thrombectomy; perfusion; anterior circulation; patient selection; endovascular therapy
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The performing interventional radiologist will be blinded for the result of the perfusion CT scan, except for the information where the occlusion of the major vessel is located.
  The assessor of the mRS score at 90 days (primary outcome) will be blinded for the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- best medical treatment and mechanical thrombectomy based on perfusion CT criteria (Experimental): In the experimental treatment group, mechanical thrombectomy is only performed when prespecified perfusion CT criteria are fulfilled. If not, the patient will only receive best medical treatment (intravenous fibrinolysis if applicable).
  Interventions: Device: perfusion CT
- best medical treatment and mechanical thrombectomy (No Intervention): All patients in the active control arm will receive the combination of best medical treatment (intravenous fibrinolysis if applicable) and mechanical thrombectomy, regardless of the results from the perfusion CT scan. This is the current standard of care for stroke patients arriving in hospital within 6 hours after onset.

INTERVENTIONS:
Device: perfusion CT — Patients are selected for thrombectomy based on perfusion CT criteria. When the results from the perfusion CT scan (analyzed by RAPID software) indicate a core infarct volume exceeding 70 ml in patients < 80 years or 55 ml in patients > 80 years, then treatment is limited to best medical treatment (intravenous fibrinolysis if applicable) and no mechanical thrombectomy will be performed. This is the current standard of care for patients treated more than 6 hour after onset.
  Other Names: RAPID software
  Arms: best medical treatment and mechanical thrombectomy based on perfusion CT criteria

SUMMARY:
The goal of this clinical trial is to test whether perfusion CT can be used as a selection tool in stroke patients with a major anterior circulation occlusion, to exclude patients from thrombectomy because of a predicted non-beneficial outcome, when treated within 6 hours of symptom onset.

Researchers will compare the experimental group, where mechanical thrombectomy is only performed when prespecified perfusion CT criteria are fulfilled, with the standard of care treatment group, where all patients will receive mechanical thrombectomy, to see if functional independence at 90 days is non-inferior.

DETAILED DESCRIPTION:
Ischemic stroke is a major cause of death or residual disability. It is caused by a blood clot blocking the brain arterial blood flow. Resolution of this blood clot can be achieved by intravenous injection of a blood clot resolving medication, if done within 4,5 h after the onset of complaints. Since about ten years, a supplementary treatment, known as mechanical thrombectomy, can be used to retrieve the blood clot from the brain circulation using a stent-retrieving system. This procedure requires an invasive transarterial approach and placement of tubes (catheter-systems) in the main brain supplying arteries to retrieve the clot by deploying stent-retrievers or by aspiration. After this maneuver, the blood supply of the brain is restored and the brain tissue that was at risk for infarction can recover. Mechanical thrombectomy has been proven to improve the functional independence of patients significantly, compared to best medical treatment alone, when performed within 6 hours of symptom onset (46% vs 26,5%).

Studies emerged on patients arriving late in the hospital, more than 6 h after onset, where mechanical thrombectomy was only performed on selected patients. Selection was based on perfusion CT scan results, which demonstrate infarction and surrounding tissue at risk (penumbra).

The functional independence was significantly better in patients who received mechanical thrombectomy versus those who only got best medical support.

In this trial the investigators aim to investigate whether the application of perfusion CT criteria to select or exclude patients from mechanical thrombectomy is non-inferior to mechanical thrombectomy without selection, with respect to functional independence at 90 days (mRS score of 0 to 2), in patients with an acute ischemic stroke caused by an occlusion of a major vessel in the anterior cerebral circulation, treated within 6 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Major vessel occlusion of the anterior cerebral circulation (internal carotid artery tip, middle cerebral artery or both) on CTA
* Randomised within 6h of symptom onset
* Perfusion CT scan
* ASPECTS ≥ 5
* Age ≥18 years and ≤90 years
* Subjects capable of giving informed consent, or if appropriate, subjects having an acceptable individual capable of giving consent on the subject's behalf (e.g. parent or guardian of a child under 16 years of age) within 3 days after treatment.

Exclusion Criteria:

* Occlusion of a peripheral arterial segment (M3), anterior cerebral artery or posterior circulation
* Evidence of intracranial hemorrhage on initial CT scan
* Bad functional condition before stroke (mRS >2)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional independence | 90 days
  Functional independence at 90 days, defined as a modified Rankin scale (mRS) score of 0 to 2. The mRS is the most comprehensive and widely used post stroke disability scale [0 (no symptoms) - 6 (death)].

SECONDARY OUTCOMES:
Early therapeutic response | hospital day 5-7 or at discharge (if before day 5)
  Early therapeutic response, defined as either a decrease in the National Institutes of Health Stroke Scale (NIHSS score) of ≥10 from baseline or an NIHSS score of 0 or 1 on hospital day 5-7 or at discharge (if before day 5). A score of 0 typically indicates normal function, while a higher score is indicative of higher level of impairment (maximum score is 42).
Health-related quality of life | 90 days
  Health-related quality of life (Euro-QoL 5D) at 3 months. The EQ-5D measures health gains as value-weighted time using quality-adjusted life years (QALYs). QALY scores range from 1 (perfect health) to 0 (dead).
Infarct evaluation | 24 hours (-6 hours / + 24 hours)
  Infarct evaluation on CT scan

OTHER OUTCOMES:
Mortality | 90 days
  Mortality rate
Intracranial bleeding | 90 days
  Intracranial bleeding rate

CONTACTS AND LOCATIONS:
Overall Officials: Luc Defreyne, Prof., Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: Undecided